CLINICAL TRIAL: NCT06585293
Title: Developing an LC-MS/MS Method for Measurement of Tacrolimus and Creatinine Concentration From Finger-prick Blood Collected Using the Mitra Device
Brief Title: Comparability of Fingerprick vs Venous Blood for Tacrolimus Monitoring
Status: Completed | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 24PA006
Record Dates: First submitted 2024-08-23; First posted 2024-09-05 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Immunosuppression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Mitra Microsampling Device — Microsampling tool for finger-prick blood collection

SUMMARY:
Organ transplant rejection occurs when the immune system attacks the transplanted organ. To prevent rejection, transplant-patients are given immunosuppressant drugs which can suppress the immune system from attacking the transplanted organ. Patients who have had a kidney-transplant take immunosuppressant drugs such as tacrolimus, but the dosage must be closely monitored through regular blood tests to avoid complications like organ failure and kidney damage. The current practice at Nottingham University Hospitals NHS Trust is that kidney-transplant patients being monitored for tacrolimus have regular blood samples taken by venepuncture (vein), and the samples are sent to the laboratory to be measured using liquid chromatography-tandem mass spectrometry (LC-MS/MS), a technique used in chemistry to identify and quantify substances in a sample. Patients will also often have their blood-creatinine measured to get an idea of kidney health. Visits to the GP/hospital for this type of blood collection can be disruptive to a patient's daily life and stretches resources of the NHS. An alternative blood sample collection process involves the use of a hand-held blood collecting device called a Mitra device, designed to allow patients to collect samples at home through a finger-prick and send them by post for analysis. This method is especially beneficial for those who find hospital visits challenging or venepuncture painful.

This study aims to develop an LC-MS/MS method for measurement of tacrolimus and creatinine, using finger-prick samples collected on the Mitra device. To do this, kidney-transplant patients who are having routine venepuncture to measure tacrolimus and creatinine will simultaneously have a finger-prick sample collected using the Mitra device. Both the venepuncture sample and finger-prick samples will be analysed using existing LC-MS/MS technology to determine tacrolimus and creatinine values. The LC-MS/MS analysis method for the finger-prick samples collected using the Mitra device will be optimised and then results obtained using this method will be compared to the results obtained from venepuncture-collected samples to ensure consistency of results. Agreement of results between the two analysis methods will confirm the suitability of LC-MS/MS method for the measurement of tacrolimus and creatinine using samples collected using the Mitra device.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending renal clinic who are receiving immunosuppressant treatment (tacrolimus) and require regular monitoring.

Exclusion Criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients attending renal clinic who are receiving immunosuppressant treatment (tacrolimus) and require regular monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Validation of an in-house LC-MS/MS method and L4L-Analyst quantitative software for the measurement of tacrolimus and creatinine using capillary fingerprick samples collected with a Mitra device. | 6 months
  Validation of an in-house LC-MS/MS method for the measurement of tacrolimus and creatinine using capillary fingerprick samples collected with a Mitra device to UKAS standards, in accordance with ISO 15189, for routine clinical practice.

SECONDARY OUTCOMES:
Questionnaire to assess whether the new sample collection method improves patient experience | 6 months
  Patient satisfaction questionnaire using a 5-point likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Donna M Fullerton, PhD, FRCPath, Principal Investigator — Nottingham University Hospitals NHS Trust
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marshall DJ, Kim JJ, Brand S, Bryne C, Keevil BG. Assessment of tacrolimus and creatinine concentration collected using Mitra microsampling devices. Ann Clin Biochem. 2020 Sep;57(5):389-396. doi: 10.1177/0004563220948886. Epub 2020 Aug 20. PMID 32713180

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-08-29): https://cdn.clinicaltrials.gov/large-docs/93/NCT06585293/SAP_000.pdf